CLINICAL TRIAL: NCT05868265
Title: Neoadjuvant Enfortumab Vedotin in High-Grade Urothelial Carcinoma of the Upper Urinary Tract (Including Ureter and Renal Pelvis)
Brief Title: A Study of Enfortumab Vedotin in People With Urothelial Carcinoma of the Upper Urinary Tract
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-393
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
Keywords: Enfortumab Vedotin; Upper Urinary Tract; High Grade; Radical surgery + pelvic lymph node dissection; 21-393
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: This is a single arm phase II trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enfortumab Vedotin (Experimental): All patients will receive enfortumab vedotin at 1.25 mg/kg on days 1 and 8 of 21 days cycle, for a total of three cycles, followed by radical nephroureterectomy, ureterectomy, or nephrectomy, depending on the site of the tumor and per the clinical decision of the treating urologist.
  Interventions: Drug: Enfortumab Vedotin; Procedure: Radical surgery

INTERVENTIONS:
Drug: Enfortumab Vedotin — All patients will receive enfortumab vedotin at 1.25 mg/kg on days 1 and 8 of 21 days cycle, for a total of three cycles.
Procedure: Radical surgery — Radical surgery, such as radical nephroureterectomy, nephrectomy or ureterectomy is to take place within 60 days from the last dose of treatment end of cycle 3 (i.e., cycle 3 day 22).

SUMMARY:
The purpose of this study is to find out whether the study drug, enfortumab vedotin, is an effective and safe treatment for people who have urothelial carcinoma of the upper urinary tract. Study participants will be people who are not eligible to receive or have chosen not to receive the chemotherapy drug cisplatin for treatment of their cancer. In addition, all participants will be planning on having standard surgery to remove their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high grade urothelial carcinoma of the upper tract and/or radiographically visible tumor stage T2-T4a N0/x M0 disease with positive selective urinary cytology. Hydronephrosis associated with tumor on imaging or biopsy will be considered invasive by definition. (Variant histology is acceptable if there is a predominant urothelial component. Discussion with PI strongly encouraged.) Retroperitoneal lymph nodes <15 mm in the short axis will be eligible.
* Patients who are

  o Ineligible for cisplatin based on any of the following criteria:
  * Estimated or calculated creatinine clearance ≥ 30ml/min but < 60 ml/min
  * Grade 2 or above audiometric hearing loss (per CTCAE v5.0) or
  * Declined cisplatin-based neoadjuvant chemotherapy, as documented in medical chart
* Availability of tumor specimen block, cell block or 30 unstained slides from diagnosis. Patients with fewer than 30 slides available may be enrolled after discussion with the Principal Investigator.Additional research biopsy is not required.
* Karnofsky performance status ≥ 70%.
* Medically appropriate candidate for radical surgery (nephroureterectomy, nephrectomy, or ureterectomy), as per treating Attending Urologic Oncologist
* Age ≥ 18 years.
* Required initial laboratory values:

  * Absolute neutrophil count ≥ 1.5 x 10^9 /L
  * Platelets ≥ 100 x 109 /L
  * Bilirubin ≤1.5 times the upper limit of normal (x ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN PTT/PT ≤1.5 x ULN or INR < 1.7 x ULN for patients who are not receiving therapeutic anticoagulation. Patients receiving therapeutic anticoagulation should be on a stable dose
* If patients are HIV (+) they are eligible as long as they have: cd4 >200, undetectable viral load and on HAART therapy.

Exclusion Criteria:

* Presence of metastatic disease.
* Prior treatment with systemic chemotherapy or radiotherapy for urothelial cancer of the bladder within the last 2 years. (Prior intravesical treatment such as BCG is allowed).
* Grade 2 or higher peripheral neuropathy.
* Patients with active keratitis or corneal ulcerations. Patients with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
* Patients with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Unstable angina.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction within 6 months.
* History of stroke within 6 months.
* Evidence of bleeding diathesis or coagulopathy. Therapeutic anticoagulation is permitted, but patients must be on a stable dose.
* Major surgical procedure within 28 days prior to the study. (Transurethral resection of bladder tumor is permitted)
* Serious, non-healing wound, ulcer, or bone fracture.
* Patients with active tuberculosis.
* Other prior malignancy active within the previous 2 years except for local or organ confined early stage cancer that has been definitively treated with curative intent or does not require treatment, does not require ongoing treatment, has no evidence of active disease, and has a negligible risk of recurrence and is therefore unlikely to interfere with the endpoints of the study.
* Prior treatment with enfortumab vedotin or other MMAE-based antibody-drug conjugates (ADCs).
* No known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Women who are breastfeeding or pregnant as evidenced by a positive pregnancy test within 14 days of first dose.
* Known severe (≥ Grade 3) hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20).
* Male subjects who are unwilling to use contraception during the treatment and for at least 31 weeks after the last dose of study treatment (5 half-lives of study drug plus 90 days duration of sperm turnover).
* Women of childbearing potential (WOCBP) not using a medically acceptable means of contraception throughout the study treatment and for at least 23 weeks following the last dose of study treatment (5 half-lives of study drug plus 30 days duration of ovulatory cycle).

  °WOCBP are defined as those who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopausal is defined as:
* Amenorrhea ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve pathologic complete response | up to 2 years
  The absence of residual disease on pathologic evaluation on surgical specimen following neoadjuvant enfortumab vedotin for UTUC. Pathologists will assess surgical specimens systematically using criteria agreed upon for all conventional neoadjuvant treatment based on the AJCC TNM staging system.

SECONDARY OUTCOMES:
The rate of grade 3 - 4 toxicity | up to 2 years
  according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Scot Niglio, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - University of Rochester Medical Center (Data Collection Only), Rochester, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm